CLINICAL TRIAL: NCT01349621
Title: Clinical Evaluation of Polarized Light Assisted Colposcopy
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daron Ferris, Professor, Department of Family Medicine and Obstetrics and Gynecology, Augusta University
Other Study IDs: CA156166; 1R21CA156166-01A1 (NIH)
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2012-09

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Abnormal Pap results; Colposcopy
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard and polarized light colposcopy: Standard and polarized light colposcopy

SUMMARY:
This is a prospective study to compare unpolarized (conventional) to polarized light colposcopy. Subjects will be asked to participate in the study when they arrive for their prescheduled colposcopic examination. The study doctor will use a conventional or standard colposcope to perform the examination. His/her impression of the exam will be noted and if necessary a biopsy specimen will be obtained. The study doctor will then perform a colposcopy using a polarized light. His/her impression of the exam will be noted and a biopsy specimen will be obtained if necessary.

This study is designed to test the hypothesis that polarized light colposcopy is more sensitive and more specific than standard, un-polarized light colposcopy.

DETAILED DESCRIPTION:
Women scheduled for a colposcopic examination at GRU or CerviCusco were asked to participate in the study. Interested patients read and signed an IRB-approved Informed Consent Document (ICD) that described the study and their potential involvement. The study coordinator read and or translated the ICD to women who spoke languages other than English or Spanish (i.e. Quechua).

Pertinent disease specific demographic information was collected from each patient. Following insertion of a vaginal speculum and a one minute application of 5% acetic acid, polarized and non-polarized high resolution digital RGB images were taken of the ectocervix. Thereafter, non-polarized light colposcopy was performed as standard of care. The colposcopist derived a colposcopic impression and indicated whether a biopsy was necessary. So as not to compromise the next examination, Lugol's Iodine was not applied. Then, a polarized light colposcopy was performed. As before, the colposcopist derived an impression, indicated whether a biopsy was necessary and annotated the site of pending biopsy. Then if indicated, a minimum of one cervical biopsy was obtained from the area(s) representing the most severe colopscopic changes as seen during the non-polarized exam. The exact biopsy site was annotated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female, 18 years or older
* Subject has previously detected abnormal cervical cytology or other indication for colposcopy
* Subject fully understands study procedures, alternative treatments available, the risks involved with the study, and voluntarily agrees to participate by giving written informed consent

Exclusion Criteria:

* Subject is pregnant or may be pregnant
* Subject has known allergy to acetic acid
* Subject has thrombocytopenia or other coagulation disorder that would contraindicate obtaining multiple cervical biopsies
* Subject is concurrently enrolled in clinical studies of investigational agents or studies involving collection of cervical specimens
* Subject has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate
* Subject has clinical evidence of gross purulent cervicitis
* Subject has a recent history of acute cervicitis
* Subject does not have an intact cervix uteri or has more than one cervix uteri

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women with a previously detected abnormal cervical cytology or other indication for colposcopy
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To determine whether polarized light increases the sensitivity and specificity over unpolarized light, the area under a receiver operating characteristic curve (AROC) will be calculated. | 8-10 months
  We will examine 300 women scheduled for colposcopy using unpolarized and polarized light. To determine whether polarized light increases the sensitivity and specificity over unpolarized light, the area under a receiver operating characteristic curve (AROC) will be calculated. We anticipate that it will take approximately 8-10 months to enroll 300 subjects.

SECONDARY OUTCOMES:
We will determine the differences in the severity of cervical neoplasia between biopsies taken using polarized and unpolarized light using a Bowker's test of symmetry. | 8-10 months
  Test the hypothesis that rates of cervical neoplasia severity detected by polarized colposcopy are greater and unpolarized colposcopy.

CONTACTS AND LOCATIONS:
Overall Officials: Daron Ferris, MD, Principal Investigator — Geogia Health Sciences University
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States